CLINICAL TRIAL: NCT05101772
Title: Multicenter, Randomized, Self-matched Design, Positive Control, Non-inferiority Clinical Study of 25G and 22G Puncture Needles in Solid or Submucosal Pancreatic Masses
Brief Title: 25G and 22G Puncture Needles
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HS-2894
Record Dates: First submitted 2021-09-18; First posted 2021-11-01 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-09

CONDITIONS: Submucosal Tumor; Pancreas Tumor
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Pancreatic or submucosal tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The screened patients were randomly assigned 25G puncture needles and 22G puncture needles in a 1;1 ratio, based on the computer-generated random order, before receiving an ultrasound endoscope puncture. Each puncture needle puncture lesions 2 needles, the same type of puncture needle tissue samples taken in the same tissue pathology bottle, all tissues after the completion of the necessary cytological smears, are placed in the Formalin solution to send tissue pathology, pathologists do not know the order of distribution of 2 puncture needles to evaluate the tissue results, all pathology results are reported by the hospital pathology center, audit.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of real pancreatic swelling or submuscular swelling;
* Patients need to be guided by ultrasound endoscopy under the guidance of puncture to eliminate malignant lesions or clear lesions;
* Fully communicate before surgery, understand the risks and benefits of endoscopic operation, and sign an informed consent form.

Exclusion Criteria:

* There are endoscopic operation contraindications, including abnormal blood clotting, or long-term oral anticoagulant antiplatelet drugs, can not guarantee INR < 1.5, or platelets less than 5 x 10 x 9 / L;
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects were 18 years of age or older (inclusive) who were clinically diagnosed with solid pancreatic masses or submucosal masses and required endoscopic ultrasound-guided puncture examination. Seventy-three subjects are planned to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Estimated)
Dates: Start 2021-09-24 (Actual); Primary Completion 2022-04-24 (Estimated); Study Completion 2022-05-24 (Estimated)

PRIMARY OUTCOMES:
The acquisition rate of the core tissue sample | One week
  A core tissue sample is defined as a sample with an histological structure that is fully used for tissue evaluation of target lesions.

SECONDARY OUTCOMES:
The length of the tissue strip | One week
  The quality of tissue samples obtained by puncture is assessed by the pathologist, whether intact tissue structure is preserved, and the length of tissue strips
the technical success rate 、the success rate of immunogrouping dyeing and the retention of the organizational structure | One week
  The quality of tissue samples obtained by punctures is evaluated by pathologists, technical success means that puncture 2 needles can obtain sufficient tissue samples for analysis to be evaluated by endoscopy.
the incidence of adverse events and the incidence of device defects | one week
  Adverse events refer to adverse medical events that occur in the course of research, including punctured complications such as bleeding, abdominal pain, infection, pancreatitis, etc. throughout the study process.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China